CLINICAL TRIAL: NCT05543382
Title: Cycling Study With the Axonics System
Status: Terminated | Type: Observational
Why Stopped: Sponsor decision not to pursue additional sites and enrollments for this study.
Sponsor: Axonics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 105-0095
Record Dates: First submitted 2022-08-15; First posted 2022-09-16 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Overactive Bladder Syndrome; Urinary Urge Incontinence; Sacral Neuromodulation
MeSH Terms: conditions — Urinary Incontinence, Urge

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Implanted group: This group will be participants with urinary urge incontinence (UUI) who have been previously implanted with an Axonics System and are satisfied with therapy
  Interventions: Device: Axonics System
- De Novo group: This group will be participants who are newly implanted with an Axonics System.
  Interventions: Device: Axonics System

INTERVENTIONS:
Device: Axonics System — The Axonics System will be implanted as standard care

SUMMARY:
A prospective, multi-center, study comparing continuous sacral neuromodulation (SNM) stimulation to daily cyclic stimulation of 2 hours "on" and 22 hours "off" using the Axonics System.

DETAILED DESCRIPTION:
After consent is provided, the required visits are at Baseline, Day 0, 1-Month, and 3-Month. At the follow-up visits, a bladder diary is reviewed, symptoms are assessed, the PGI-I questionnaire is completed, and cyclic stimulation hours may be changed.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who are ≥ 21 years at the time of consent
2. Has a primary indication of UUI (participants with a secondary indication of UF or FI may also be enrolled)
3. Has a diagnosis of UUI for greater than or equal to 6 months prior to the date of consent
4. UUI episodes:

   1. For currently implanted participants (Group A), they must be considered therapy responders with a >50% reduction in UUI episodes (based on their original baseline diaries) and satisfied with their SNM therapy
   2. For de novo candidates (Group B), they must have completed a successful PNE documented with a >50% reduction in UUI episodes on a 3-day diary (a diary must exist within a medical record or equivalent)
5. Willing and capable of providing informed consent
6. Agrees to return to the site for all study visits
7. Fluent (able to speak and read) in English

Exclusion Criteria:

1. Any participant that the study Investigator deems to be a poor candidate who is unable to complete a 72-hour bladder diary or will be non-compliant for study visits
2. Diagnosis of urinary retention
3. Surgical treatment for stress incontinence (e.g. sling, Burch), and/or pelvic organ prolapse in the past 3 months or recommended or planned within 3 months from the time of consent
4. Changes to current regimen of medications that could impact bladder function within 4 weeks prior to consent
5. Current urinary tract mechanical obstruction (e.g., benign prostatic enlargement or urethral stricture)
6. Current symptomatic urinary tract infection (UTI)
7. A patient who early discontinued from the ARTISTRY registry
8. A female with a positive urine pregnancy test
9. A female who is breastfeeding

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The sample size will include 60 de novo participants with UUI, or currently implanted participants with UUI. Participants may be implanted with either the rechargeable or recharge-free Axonics Systems.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2022-08-09 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2024-12-29 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of daily cyclic stimulation of 2 hours "on" and 22 hours "off" in reducing UUI episodes by > 50% in newly implanted participants, or maintenance of efficacy in currently implanted participants with an implanted Axonics System | 3 months
  Comparison of UUI episodes on a 3-day bladder diary at 3 months as compared to baseline UUI episodes

SECONDARY OUTCOMES:
To evaluate patient satisfaction with cyclic stimulation | 3 months
  Analysis of the Patient Global Impression of Improvement (PGI-I) scale. This scale evaluates the post-operative condition. The PGI-I has 1 question with 7 possible answers ranging from "very much better" (score of 1) to "very much worse" (score of 7).

CONTACTS AND LOCATIONS:
Overall Officials: Karen Noblett, MD, Study Director — Axonics, Inc.
Locations (6):
- United States (6):
  - The Florida Bladder Institute, Naples, Florida
  - LSU Health, New Orleans, Louisiana
  - University Hospitals-Cleveland Medical Center, Cleveland, Ohio
  - Urologic Specialists Oklahoma, Tulsa, Oklahoma
  - The Female Pelvic Health Center, Newton, Pennsylvania
  - Center for Pelvic Health, Franklin, Tennessee

IPD SHARING:
Plan to Share IPD: No